CLINICAL TRIAL: NCT05678465
Title: MEsh FIxation in Laparoendoscopic Repair of Large M3 Inguinal Hernias - Multicenter, Double-blinded, Randomized Controlled Trial.
Brief Title: MEsh FIxation in Laparoendoscopic Repair of Large M3 Inguinal Hernias
Acronym: MEFI
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Swissmed Hospital (Other)
Collaborators: Klinika Chirurgii Ogólnej, Onkologicznej i Endokrynologicznej Szpitala Zespolonego w Kielcach (Unknown); Oddział Chirurgii Ogólnej MCM Jonscher w Łodzi (Unknown); Oddział Chirurgii Ogólnej i Onkologicznej Szpitala w Wejherowie (Unknown); Klinika Chirurgii Ogólnej i Onkologicznej UM w Łodzi (Unknown); Oddział Chirurgii Ogólnej, Małoinwazyjnej i Wieku Podeszłego Miejskiego Szpitala Zespolonego w Olsztynie (Unknown); Oddział Chirurgii Ogólnej Regionalnego Centrum Zdrowia w Lubinie (Unknown); Klinika Chirurgii Ogólnej, Wojskowy Instytut Medycyny Lotniczej w Warszawie (Unknown); Oddział Chirurgii Ogólnej, SPOZ w Siedlcach (Unknown); Oddział Chirurgii Ogólnej Szpitala w Puszczykowie (Unknown); Oddział Chirurgii Ogólnej z Pododdziałem Urazowo-Ortopedycznym Szpitala w Szczytnie (Unknown); Oddział Chirurgiczny Ogólny, Wojewódzki Szpital Specjalistyczny w Częstochowie (Unknown)
Responsible Party: Principal Investigator, Mateusz Zamkowski, MD, PhD, Swissmed Hospital
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: MEFI TRIAL
Record Dates: First submitted 2022-12-26; First posted 2023-01-10 (Actual); Last update posted 2024-10-15 (Actual); Status verified 2024-10

CONDITIONS: Hernia, Inguinal; Hernia, Direct Inguinal
Keywords: hernia; tapp; inguinal hernia; laparoendscopic repair; groin hernia; mesh
MeSH Terms: conditions — Hernia, Inguinal; Hernia

STUDY DESIGN:
Intervention Model Description: Patients in both arms will recieve intervention. First arm (mesh + fixation) serves also as control. Patients in second arm will be operated with mesh without fixation.
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: Double-blinded (surgeon/patient)
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- FIXATION (Experimental): Lightweight macroporous mesh at least 15x10cm will be placed in preperitoneal space and fixated with use of histoacryl glue.
  Mesh - B Braun® Optilene Mesh® or BD® SoftMesh® Glue - Histoacryl® LapFix
  Interventions: Procedure: Fixation of the mesh
- NON-FIXATION (Experimental): Standard, 3-D, anatomical mesh will be placed in preperitoneal space without the use of fixating materials.
  Mesh - BD® 3D Max® Mesh or Medtronic® Dextile Anatomical Mesh®
  Interventions: Procedure: Non-fixation of the mesh

INTERVENTIONS:
Procedure: Non-fixation of the mesh — 3D-shaped, anatomical, standard, polypropylene mesh without fixation.
  Other Names: 3D Max Mesh (BD); Dextile Anatomical Mesh (Medtronic)
  Arms: NON-FIXATION
Procedure: Fixation of the mesh — Glue fixation of lightweight, macroporous, polypropylene mesh.
  Other Names: B Braun Optilene Mesh; BD SoftMesh
  Arms: FIXATION

SUMMARY:
The goal of this Multicenter Clinical Trial is to verify the hypothesis that non-fixation of the 3-D anatomical mesh (Dextile Anatomical Mesh or 3D Max Mesh) is non-inferior in terms of recurrence compared to fixation of lightweight, macroporous meshes in laparoendoscopic repairs of large M3 inguinal hernias.

DETAILED DESCRIPTION:
INTRODUCTION International guidelines of groin hernia treatment strongly recommends to fixate the mesh in case of large M3 medial defects during laparoendoscopic approach (TAPP / TEP). Main purpose of fixation is to decrease recurrence rate which is alarmingly high in case of those defects. Recommendation was based on analysis of large German database (Herniamed). However, deeper look into those findings shows that most of TAPP and TEP procedures were performed with the use of lightweight, flat, macroporous meshes. In 2022 multidisciplinary team consisting of hernia surgeons and scientists from universities of technology conducted an experimental study with the use of 3d groin model to confirm or deny the hypothesis that fixation is not necessary in above cases. Study was conducted with the use of all 3-D anatomical meshes available on Polish market, as well as with flat, macroporous implants. Experiment showed that large, rigid and anatomically shaped meshes are able to maintain its position in groin without need of fixation. To confirm experimental results we decided to conduct large, multicentre, clinical study to evaluate necessity of mesh fixation of large, spatial, standard polypropylene implants.

STUDY HYPOTHESIS Non-fixation of spatial, standard polypropylene meshes is non-inferior as compared to fixation of flat, polypropylene lightweight meshes during TAPP / TEP procedures.

MATERIALS AND METHODS 11 large surgery centres in Poland having proficiency in laparoendoscopic groin hernia repairs (performing at least 80 TAPP/TEP a year) were recruited for this study. Before recruiting patients a two day "bootcamp" meeting was planned. Each centre designated one surgeon responsible for conducing the trial in its hospital and sent him/her to meeting. Recurrence rate in 12-month follow-up was set as a primary endpoint. Pain sensation (assessed with VAS scale) was made a secondary endpoint. Statistical analysis was performed by experts to adjust the sample sizes. The trial was planned as non-inferiority study with test power = 80%, p-value = 0,05 and threshold for clinical significance = 8%. Percentage loss was assumed at 10%. Recurrence rate was assumed 4% based on literature. Based on those assumptions minimal sample size in both arms was calculated at 83-102. Inclusion criteria: elective groin hernia repair, age > 18 years, male and female patients can participate, M3 or M3+L1-3 (EHS classification) groin hernia confirmed during surgery, eligibility to laparoendoscopic repair, written informed consent. Exclusion criteria: age <18 years, emergency surgery (incarcerated hernia), contaminated surgical field, extremely large scrotal hernia with the need of other forms of prevention of ACS (preoperative botox injection, bowel resection etc.) First arm (control group) will consist of patients repaired with the use of flat, macroporous, lightweight mesh fixated with histoacryl glue. Second arm will consist of patients repaired with the use of anatomically shaped, large, standard, polypropylene mesh (Dextile Anatomical Mesh - MEDTRONIC or 3D Max Mesh - BD) without the use of fixation material.

As M3 hernias are difficult to diagnose before the surgery, all patients planned for laparoendscopic repairs will be asked to participate in trial. During the surgery, when the defect size is measured, patient will be fully included in the study. After dissection of preperitoneal space (and establishing crucial checkpoints), surgeon will open envelope and find out the technique he will have to perform. Patients won't be aware of the method used during surgery. Unblinding will take place at the end of the trial. Pain will be measured during the hospital stay and then 7-days, 3-months and 12-months after surgery (VAS Scale). Follow up will be performed by Medical Assistant via phone call (also blinded to the method used). If any doubts occur, patient will be asked to come to ambulatory visit.

PREDICTED OUTCOMES Based on experimental study published in Surgical Endoscopy (Zamkowski et al., 2022) and own experience, we believe that recurrence rate in both arms will be on the same level. Those outcomes will be a strong argument for amending the guidelines in terms of mesh fixation. It would show that mesh fixation is not necessary if the proper, spatial mesh is used.

ELIGIBILITY:
Inclusion Criteria:

* elective groin hernia repair,
* M3 or M3+L1-3 (EHS classification) groin hernia confirmed during surgery
* eligibility to laparoendoscopic repair
* written informed consent

Exclusion Criteria:

* emergency surgery (incarcerated hernia)
* contaminated surgical field
* recurrent hernia
* extremely large scrotal hernia with the need of other forms of prevention of Abdominal Compartment Syndrome (botox injection, preoperative progressive pneumoperitoneum - PPP, bowel resection etc.)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 204 (Actual)
Dates: Start 2023-02-01 (Actual); Primary Completion 2023-11-30 (Actual); Study Completion 2024-10-12 (Actual)

PRIMARY OUTCOMES:
Reccurence Rate | 12-months
  Reccurence in 1 year after surgery

OTHER OUTCOMES:
Pain score | 7-days, 3-months, 12-months
  Pain sensation using Pain Visual Analog Scale (VAS)
Other complications | 7-days, 3-months, 12-months
  Other surgical complications (seroma, hematoma, surgical site infections - SSI etc.)

CONTACTS AND LOCATIONS:
Overall Officials: Mateusz Zamkowski, MD, PhD, Study Chair — Swissmed Hospital; Maciej Śmietański, Prof., Study Director — Swissmed Hospital
Locations (1):
- Swissmed Hospital, Gdansk, Poland

IPD SHARING:
Plan to Share IPD: Yes
Data will be availble in English on a reasonable request.
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: Data will be availble in English on a reasonable request.
Access Criteria: Access to trial IPD can be requested by qualified researchers engaging in independent scientific research, and will be provided following review and approval of a research proposal and Statistical Analysis Plan (SAP) and execution of a Data Sharing Agreement (DSA). For more information or to submit a request, please contact.

REFERENCES:
- [Background] Zamkowski M, Tomaszewska A, Lubowiecka I, Karbowski K, Smietanski M. Is mesh fixation necessary in laparoendoscopic techniques for M3 inguinal defects? An experimental study. Surg Endosc. 2023 Mar;37(3):1781-1788. doi: 10.1007/s00464-022-09699-5. Epub 2022 Oct 13. PMID 36229552
- [Background] HerniaSurge Group. International guidelines for groin hernia management. Hernia. 2018 Feb;22(1):1-165. doi: 10.1007/s10029-017-1668-x. Epub 2018 Jan 12. PMID 29330835
- [Background] Mayer F, Niebuhr H, Lechner M, Dinnewitzer A, Kohler G, Hukauf M, Fortelny RH, Bittner R, Kockerling F. When is mesh fixation in TAPP-repair of primary inguinal hernia repair necessary? The register-based analysis of 11,230 cases. Surg Endosc. 2016 Oct;30(10):4363-71. doi: 10.1007/s00464-016-4754-8. Epub 2016 Feb 17. PMID 26886454
- [Background] Novik B, Sandblom G, Ansorge C, Thorell A. Association of Mesh and Fixation Options with Reoperation Risk after Laparoscopic Groin Hernia Surgery: A Swedish Hernia Registry Study of 25,190 Totally Extraperitoneal and Transabdominal Preperitoneal Repairs. J Am Coll Surg. 2022 Mar 1;234(3):311-325. doi: 10.1097/XCS.0000000000000060. PMID 35213495
- [Derived] Zamkowski M, Smietanski M. MEsh FIxation in Laparoendsocopic Repair of Large M3 inguinal hernias: multicenter, double-blinded, randomized controlled trial-study protocol for a MEFI Trial. Trials. 2023 Sep 5;24(1):572. doi: 10.1186/s13063-023-07601-9. PMID 37670376